Clinical Study of the WoundCare360 SiteSeal Adjunctive Compression Device Following Interventional Endovascular Procedures – NCT03234894

**Informed Consent Form:** 

Document Date: April 23, 2015



Protocol: 15-003 April23, 2015

| Woundcare 360 |
|---------------------------|
| 10900 S. Clay Blair Blvd. |
| Olathe, KS 66061 |

| Olathe, KS 66061 | | | |
|-------------------|-------------|----------------|------------|
| Patient ID: | | DOB (mm/dd/yyy | <b>y</b> ] |
| Patient Initials: | Visit Date: | _(mm/dd/yyyy) | |

#### Eligibility

Please enter responses in space provided.

- 1. Has this patient met all eligibility criteria according to the protocol?
  - a. YES NO

Inclusion Criteria All must be "YES" to qualify.

| Is patient's age between19 to 90? | YES | NO |
|---|---|---|
| Has patient given written informed consent for participation prior | YES | NO |
| to the procedure? | | |
| Is this procedure an interventional procedure? | YES | NO |
| Is patient willing to undergo all study procedures and adhere to | YES | NO |
| data collection and follow-up requirements? | | |
| Is patient a candidate for elective, non-emergent cardiac or | YES | NO |
| peripheral vascular catheterization from the femoral artery | | |
| approach? | | |
| Is patient willing to have a pre/post procedure ultrasound? | YES | NO |

### Exclusion Criteria All must be "NO" to qualify.

| Is patient's age <19 years? | YES | NO |
|-----------------------------------------------------------------|-----|----|
| Is patient's age > 90 years? | YES | NO |
| Did the patient receive GP IIb/IIIa inhibitors? | YES | NO |
| Is patient able to provide written informed consent on his/her | YES | NO |
| own behalf? | | |
| Is patient unable or unwilling to adhere to data collection and | YES | NO |
| follow-up requirements? | | |
| Is the procedure emergency PCI? | YES | NO |
| Is the patient on dialysis? | YES | NO |
| Does the patient have a known diagnosis of fibromyalgia? | YES | NO |



Protocol: 15-003 April23, 2015

Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061

| Patient ID: | | DOB | (mm/dd/yyyy) |
|-------------------|-------------|--------------|--------------|
| Patient Initials: | Visit Date: | (mm/dd/yyyy) | |

| Does the patient have acute coronary syndrome (i.e., unstable angina or myocardial infarction) $\leq 48$ hours before this catheterization procedure? | YES | NO |
|---|---|---|
| Was the patient's systolic blood pressure < 90 mm Hg at the end of this catheterization procedure? | YES | NO |
| Is the patient immunocompromised? | YES | NO |
| Does the patient have pre- existing systemic infection or local infections at this access site? | YES | NO |
| Is the patient known or suspected to be pregnant, or is lactating? | YES | NO |
| Has the patient undergone prior or recent use of an intra- aortic balloon pump through the arterial access site? | YES | NO |
| Has the patient undergone prior vascular closure device use in the ipsilateral common femoral artery $\leq 30$ days before this catheterization procedure? | YES | NO |
| Has the patient undergone prior use of manual or mechanical compression for closure in the ipsilateral common femoral artery ≤ 30 days before this catheterization procedure? | YES | NO |
| Did the patient require a re- puncture at a site previously punctured within 48 hours of this catheterization procedure? | YES | NO |
| Did the patient have an antegrade puncture in this catheterization procedure? | YES | NO |
| Did the patient have a puncture site believed to be in the profunda femoris artery, superficial femoral artery, or at the bifurcation of these arteries in this catheterization procedure? | Yes | NO |
| Was the patient's puncture tract angle > 55° in this catheterization procedure? | YES | NO |
| Is the patient suspected to have experienced a femoral artery back wall puncture or who underwent > 1 femoral artery puncture during this catheterization procedure? | YES | NO |



Protocol: 15-003 April23, 2015

Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061

| Patient ID: | | DOB | (mm/dd/yyyy) |
|-------------------|-------------|--------------|--------------|
| Patient Initials: | Visit Date: | (mm/dd/yyyy) | |

| Does the patient have significant anemia (hemoglobin < 10 g/dL, Hct < 30%)? | YES | NO |
|---|---|---|
| Does the patient have a known bleeding disorder, including thrombocytopenia (platelet count < 100,000 cells/µL), thrombasthenia, hemophilia, or von Willebrand's disease? | YES | NO |
| Did the patient have systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg at the end of this catheterization procedure, unless systolic and/or diastolic pressure was lowered by pharmacological agents prior to the end of this catheterization procedure? | YES | NO |
| Did the patient have a baseline INR > 1.5 (e.g., on warfarin therapy)? | YES | NO |
| Was the patient's ACT > 300 seconds at the end of this catheterization procedure? | YES | NO |
| Did the patient undergo administration of low molecular weight heparin (LMWH) within 8 hours of this catheterization procedure? | YES | NO |
| Is continued heparin or other anticoagulant/antiplatelet therapy planned for this patient (with the exception of glycoprotein IIb/IIIa inhibitor therapy) during the first few hours following this catheterization procedure? | YES | NO |
| Did the patient have a complication or complications at the femoral artery access site during the catheterization procedure including bleeding, hematoma, intraluminal thrombus, pseudoaneurysm, or arteriovenous fistula? | YES | NO |
| Does the patient have an ipsilateral or bilateral lower extremity amputation(s)? | YES | NO |
| Is the patient known to require extended hospitalization (e.g., patient is undergoing cardiac surgery)? | YES | NO |



Signature

Protocol: 15-003 April23, 2015 Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061 DOB \_\_\_\_\_(mm/dd/yyyy) Patient ID: \_\_\_\_\_ Patient Initials: \_\_\_\_ Visit Date: \_\_\_\_\_\_ (mm/dd/yyyy) Does the patient have a planned endovascular procedure within YES NO the next 30 days after this catheterization procedure? NO Is the patient currently participating in another investigational YES study that has not concluded the follow- up period? Has the patient already participated in this IDE study? YES NO Is it known that the patient cannot adhere to or complete the YES NO study for any reason including but not limited to geographical residence or life- threatening disease?

Date (mm/dd/yyyy)



7. Systolic blood pressure

a. \_\_\_\_\_ mm Hg

Protocol: 15-003 April23, 2015 Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061 DOB \_\_\_\_\_(mm/dd/yyyy) Patient ID: \_\_\_\_\_ Patient Initials: \_\_\_\_\_ Visit Date: \_\_\_\_\_ (mm/dd/yyyy) Demographics 1. Date of Birth: \_\_\_\_\_\_ (dd/mm/yyyy) 2. Gender: MALE FEMALE 3. Race a. Caucasian b. Hispanic c. Asian d. Black e. Other 4. Height: \_\_\_\_\_ (ft/inches) 5. Weight: \_\_\_\_\_ (lbs) 6. BMI: \_\_\_\_\_ Procedure-Related Data 1. Procedure Type: a. CARDIAC PERIPHERAL VASCULAR 2. Access Site Location a. RIGHT LEFT 3. Size of the introducer sheath: a. \_\_\_\_Fr. 4. Intra-procedure anticoagulants: 5. Intra-procedure antiplatelet agents: 6. Previous arterial puncture site in the ipsilateral common femoral artery >30days before this catheterization procedure: a. YES NO



Protocol: 15-003 April23, 2015

| woundcare 360<br>10900 S. Clay Blair Blvd.<br>Olathe, KS 66061 | | | |
|---|---|---|---|
| Patient ID: | | DOB | (mm/dd/yyyy) |
| Patient Initials: | _ Visit Date: | (mm/dd/yyy | y) |
| a<br>11. Pre-procedural a<br>a<br>12. Pre-procedure a<br>a<br>13. Post-procedural | mm Hg ial disease: g time (ACT) at the e seconds anticoagulants: ntiplatelet agents (in | | · |
| PREVIOUS DIAGNOSTIO | C/INTERVENTIONAL | ENDOVASCULAR PRO | CEDURES |



pain

Protocol: 15-003 April23, 2015 Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061 Patient ID: \_\_\_\_\_ DOB \_\_\_\_\_(mm/dd/yyyy) Visit Date: \_\_\_\_\_(mm/dd/yyyy) Patient Initials: \_\_\_\_\_ Catheterization Procedure Data 1. Procedure Date: \_\_\_\_\_\_ (mm/dd/yyyy) 2. Pre-procedure Duplex Ultrasound? a. YES NO 3. Procedure Start Time: a. \_\_\_\_\_(24hour) 4. Procedure End Time: a. \_\_\_\_\_(24hour) 5. Post procedure Duplex Ultrasound? a. YES NO 6. Time of SiteSeal removal: a. \_\_\_\_\_(24hour) 7. Calculated time to deploy device without visible bleeding at the access site (TTH): a. 8. Time of first standing & walking 20ft without evidence of arterial re-bleeding from the access site (TTA): a. (24hour) 9. Calculated Time To Ambulation (TTA): a. (24hour) 10. Adverse events: a. YES NO 11. Patient Discomfort: a. Patient discomfort @ discharge from the catheterization lab: i. Patient comfort level (1-10) with 10 being intense b. Patient discomfort @ 24 hours after this procedure: i. \_\_\_\_\_ Patient comfort level (1-10) with 10 being intense



Protocol: 15-003 April23, 2015

Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061

| Olathe, KS 66061 | | | |
|-------------------|-------------|---------------|--------------|
| Patient ID: | | DOB | (mm/dd/yyyy) |
| Patient Initials: | Visit Date: | _(mm/dd/yyyy) | |

#### Primary Post Procedure Endpoints

#### 1. Nerve Puncture

- a. Was there an involuntary leg muscle contraction and an auditory response at the time of placing the device?
  - i. YES NO

#### 2. Femoral Artery Laceration

- a. Was there common femoral artery laceration (or needle penetration) with resultant bleeding or hematoma > 6 cm diameter?
  - i. YES NO

#### Secondary Endpoints

#### Major Complications @ 30day follow-up

- 1. Vascular repair or the need for vascular repair (via surgery, ultrasound-guided compression, transcatheter embolization, or stent-graft) Y N
- 2. Access site-related bleeding requiring transfusion Y N
- 3. Any new ipsilateral lower extremity ischemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram Y N
- 4. Surgery or the need for surgery for access site-related nerve injury Y N
- 5. Permanent (lasting > 30 days) access site-related nerve injury Y N
- Access site-related infection requiring intravenous antibiotics and/or extended hospitalization – Y N



Protocol: 15-003 April23, 2015

Woundcare 360 10900 S. Clay Blair Blvd. Olathe, KS 66061

| Olathe, KS 66061 | | | |
|-------------------|-------------|--------------|--------------|
| Patient ID: | | DOB | (mm/dd/yyyy) |
| Patient Initials: | Visit Date: | (mm/dd/yyyy) | |

#### Minor Complications @ 30day Follow-up

- 1. Non-treated pseudoaneurysm documented by ultrasound Y N
- 2. Non-treated arteriovenous (AV) fistula documented by ultrasound Y N
- 3. Pseudoaneurysm treated with ultrasound-guided thrombin injection or ultrasound-guided fibrin adhesive injection Y N
- 4. Access site hematoma greater than or equal to 6 cm Y N
- 5. Access site-related bleeding requiring greater than 30 minutes to achieve hemostasis Y N
- 6. Late (following hospital discharge) access site-related bleeding Y N
- 7. Ipsilateral lower extremity arterial emboli Y N
- 8. Transient loss of ipsilateral lower extremity pulse Y N
- 9. Ipsilateral deep vein thrombosis Y N
- 10. Access site-related vessel laceration Y N
- 11. Transient access site-related nerve injury Y N
- 12. Access site wound dehiscence Y N
- 13. Localized access site infection treated with intramuscular or oral antibiotics Y N